CLINICAL TRIAL: NCT04139928
Title: Bioavailability of Single-dose Magnesium Salts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Think Healthy Group, Inc. (Network)
Collaborators: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: THG-IU-MG-1
Record Dates: First submitted 2019-10-23; First posted 2019-10-25 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Bioavailability
Keywords: Magnesium
MeSH Terms: interventions — magnesium citrate; Magnesium Oxide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Picometer-ionic form of magnesium chloride (Experimental)
  Interventions: Dietary Supplement: Picometer-ionic form of magnesium chloride
- Magnesium citrate or magnesium oxide (Active Comparator)
  Interventions: Dietary Supplement: Magnesium citrate or magnesium oxide
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Picometer-ionic form of magnesium chloride — Single-dose (300 mg) of the picometer-ionic form of magnesium chloride
  Arms: Picometer-ionic form of magnesium chloride
Dietary Supplement: Magnesium citrate or magnesium oxide — Single-dose (300 mg) of magnesium citrate or magnesium oxide
  Arms: Magnesium citrate or magnesium oxide
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Magnesium plays a role in an array of critical body functions, controls normal adenosine triphosphate function, the metabolism of glucose, and cardiac muscle function, as well as the maintenance of cell membrane function. Low magnesium intakes and blood levels have been associated with a number of chronic diseases including hypertension, type 2 diabetes, metabolic syndrome, vascular disease, osteoporosis, and colon cancer. Magnesium deficiency is common. In the U.S. population, nearly 4% of men and 7% of women have hypomagnesemia (typically defined as a serum concentration <0.75 mmol/L, or < 17mg/L), which has been previously shown to be associated with an increased risk of all-cause mortality after 30 years of follow-up. In addition, hypomagnesemia is seen in approximately 11% of hospitalized patients and 52% of patients in coronary care units. Approximately half of the U.S. population does not currently reach the estimated average requirement (EAR) for magnesium from food. Yet magnesium deficiency is often overlooked.

Magnesium is relatively well absorbed by the gut; oral bioavailability varies from 35 to 70% and depends on a variety of factors such as the form of the magnesium salt (organic vs. inorganic), its rate and extent of uptake from the intestine into the blood, and its transfer into tissues because magnesium is primarily an intracellular cation. The absorption rate increases when dietary intake is low. In terms of the effectiveness of oral dietary supplements, bioavailability and tolerability of various formulations are important considerations. Similar bioavailability has been demonstrated between inorganic formulations (magnesium oxide vs. magnesium chloride), however some studies have shown magnesium oxide to be less bioavailable. Diarrhea and abdominal cramping are side effects that are commonly reported from oral oral supplementation. These symptoms are thought to be due to the osmotic activity of unabsorbed salts in the intestine and colon and the stimulation of gastric motility. A new picometer-ionic form of magnesium chloride, was developed to efficiently deliver stabilized magnesium ions that are similar in size to plant magnesium. Picometer magnesium is smaller in diameter than the body's cell mineral ion channels, therefore it has the potential to be completely absorbed and not cause adverse side effects in the gastrointestinal system (e.g., diarrhea). The aim of this research is to assess the bioavailability of this new picometer-ionic form of magnesium chloride by comparing its bioavailability to that of a standard magnesium oxide and magnesium citrate supplement in healthy, adult, normotensive subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18- 65 years
2. Body mass index 18 to 35 kg/m2 , body weight ≥ 110 pounds or 50 kg
3. All race/ethnicities and both sexes, are eligible.
4. Normal blood pressure (BP) ≤ 120/80 mm Hg.

Exclusion Criteria:

1. Participant has a diagnosis of hypertension, prehypertension, diabetes, cardiovascular or other chronic disease (e.g., cancer).
2. Participant has a diagnosis of hypermagnesemia (defined as a serum concentration of > 22.8 mg/L of Magnesium) (4).
3. Participant is already taking magnesium supplementation prior to the study or taking medications that interfere with magnesium metabolism, we are providing examples in an appendix.
4. Participant has concurrent use of magnesium supplements and/or other nutrient supplements that interfere with magnesium absorption (e.g., calcium supplements) within 2-wk prior the first treatment or during the course of this study.
5. Participant has gastrointestinal disease, hepatitis, anemia, or hepatic enzyme abnormalities.
6. Women subjects are currently pregnant or trying to become pregnant.
7. Participant has a history of hospitalization for acute illness in the previous 1 month.
8. Participants who do not speak English or are unable to read or fail to comprehend the informed consent form.
9. Participants fail to complete the full medical questionnaire reviewed with them during the initial phone call (whether it be because they refuse to answer or because they don't know/understand the questions).
10. Participants who have a body weight less than 110lbs (or 50kg).
11. Participants who have donated blood within the last month, or are currently giving blood for other clinical or research purposes.
12. Participants who smoke and/or use tobacco products.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-03-24 (Actual); Study Completion 2020-04-28 (Actual)

PRIMARY OUTCOMES:
Ionized magnesium (whole blood) | 24 hours
  Ionized magnesium in whole blood is the primary outcome measure which will be measured by using a magnesium selective electrode clinical analyzer (Stat Profile Prime® Model, Prime Electrolyte System) at multiple time points following the oral doses of the magnesium supplements (MgCl vs MgO vs placebo). The time points will be -15 minutes prior to dose and post dose at 30 minutes, 1 hour, 2 hour, 3 hour, 4 hour, 6 hour, 8 hour and 24 hour.
Total magnesium in serum and urine | 24 hours
  Total magnesium in serum and urine are the secondary outcome measures which will be measured by using inductively coupled plasma-mass spectrometry (ICP-MS) at multiple time points following the oral doses of the magnesium supplements (MgCl vs MgO vs placebo). The time points for serum total magnesium will be -15 minutes prior to dose and post dose at 30 minutes, 1 hour, 2 hour, 3 hour, 4 hour, 6 hour, 8 hour and 24 hour. Complete urine collections will be obtained at pooled intervals that coincide with timing of blood draws.
Exploratory / Correlative Outcome Measures | 24 hours
  A reference range for ionized magnesium in whole blood in healthy adults will be established for the magnesium selective electrode clinical analyzer.

CONTACTS AND LOCATIONS:
Overall Officials: Taylor C. Wallace, PhD, Principal Investigator — Think Healthy Group, LLC; Nana Gletsu-Miller, PhD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ansu Baidoo VY, Thiagarajah K, Tekwe CD, Wallace TC, Gletsu-Miller N. Relationship between short-term self-reported dietary magnesium intake and whole blood ionized magnesium (iMg2+) or serum magnesium (s-Mg) concentrations. Ann Med. 2023 Dec;55(1):2195702. doi: 10.1080/07853890.2023.2195702. PMID 37036758
- [Result] Zhan J, Wallace TC, Butts SJ, Cao S, Ansu V, Spence LA, Weaver CM, Gletsu-Miller N. Circulating Ionized Magnesium as a Measure of Supplement Bioavailability: Results from a Pilot Study for Randomized Clinical Trial. Nutrients. 2020 Apr 28;12(5):1245. doi: 10.3390/nu12051245. PMID 32353962